CLINICAL TRIAL: NCT02985333
Title: Efficacy and Safety of Paclitaxel/Cyclophosphamide/Dexamethasone to Treat Patients With Relapsed or Refractory Multiple MyelomaRefractory
Brief Title: Paclitaxel,Cyclophosphamide and Dexamethasone for Relapsed or Refractory Multiple Myeloma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, wanghua, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM-2014
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2018-05-14 (Actual); Status verified 2016-12

CONDITIONS: Relapse/Refractory Multiple Myeloma
Keywords: paclitaxe,cyclophosphamide,dexamethasone, Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Paclitaxel; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): paclitaxel 175 mg/m(2) IV over 3 h d1,cyclophosphamide 200 mg/m(2) IV d1,3,5 and dexamethasone 20mg IV d1-4 in patients with relapsed or refractory MM.
  Interventions: Drug: Paclitaxel; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 170 mg/m(2) IV over 3 h d1
  Other Names: Taxol
Drug: Cyclophosphamide — Cyclophosphamide 200mgmg/m(2) IV d1,3,5
  Other Names: cytoxan
Drug: Dexamethasone — Dexamethasone 20mg iv d1-4
  Other Names: hexadecadrol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of paclitaxel in combination with cyclophosphamide and dexamethasone in chinese patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Treatment for relapsed/refractory multiple myeloma (MM)remains a crucial challenge.The investigators have previously shown that the combination of paclitaxel and cyclophosphamide acts synergistically to induce apoptosis of myeloma cells in vitro. Based on these preclinical studies, the investigators initiated a phase II clinical trial of paclitaxel 175 mg/m(2) IV over 3 h d1 combined with cyclophosphamide 200 mg/m(2) IV over 30-60 min d1,3,5 and dexamethasone 20mg IV over 30-60 min d1-4 in patients with relapsed or refractory MM. This regimen was administered every four weeks for a total of six cycles

ELIGIBILITY:
Inclusion Criteria:

* Patient has a previous diagnosis of multiple myeloma
* Patient requires retreatment for multiple myeloma
* Subject has measurable disease as defined by > 0.5 g/dL serum monoclonal protein, >10 mg/dL involved serum free light chain (either kappa or lambda) provided that the serum free light chain ratio is abnormal, >0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s) of at least 1cm in greatest dimension as measured by either CT scanning or MRI
* Subject has a Karnofsky performance status ≥60% (>50% if due to bony involvement of myeloma (see Appendix IV)
* Subject has a life expectancy ≥ 3 months
* Subjects must meet the following laboratory parameters:

Absolute neutrophil count (ANC) ≥750 cells/mm3 (1.0 x 109/L) Hemoglobin ≥ 7 g/dL Platelet count ≥ 75,000/mm3 (30 x 109/L if extensive bone marrow infiltration) Serum SGOT/AST <3.0 x upper limits of normal (ULN) Serum SGPT/ALT <3.0 x upper limits of normal (ULN) Serum total bilirubin <2.0 mg/dL (34 µmol/L) Creatinine clearance ≥ 45 cc/min

Exclusion Criteria:

* Subject has immeasurable MM (no measurable monoclonal protein, free light chains in blood or urine, or measureable plasmacytoma on radiologic scanning)
* Subject has a prior history of other malignancies unless disease-free for ≥ 5 years, except for basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix or breast, or localized prostate cancer with Gleason score < 7 with stable prostate specific antigen (PSA) levels
* Subject has had myocardial infarction within 6 months prior to enrollment, or NYHA (New York Hospital Association) Class III or IV heart failure (see Appendix VI), Ejection Fraction < 35%, uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Female subject who is pregnant or lactating
* Subject has known HIV infection
* Subject has known active hepatitis B or hepatitis C infection
* Subject has active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program
* Subject is unable to reliably take oral medications
* Subject has known hypersensitivity to dexamethasone,cyclophosphamide,paclitaxel
* Subject has a history of thromboembolic event within the past 4 weeks prior to enrollment
* Subject has any clinically significant medical or psychiatric disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 30 months
  ORR is defined as the proportion of patients with CR, nCR or partial response (PR) based on modified EBMT criteria per investigator assessment

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | 30 months
  PFS, defined as time from first dose of study treatment to progression or death due to any cause, as assessed by investigator
Overall survival (OS) | 30 months
  OS, defined as time from first dose of study treatment to death
Safety of combination therapy assessed using the National Cancer institute-Common Toxicology Criteria (NCI-CTC) grade scale for AEs and Lab assessments | 30 months
  Safety of combination therapy as assessed by toxicity, which will be assessed using the National Cancer Institute-Common Toxicology Criteria (NCI-CTC) grading scale for Adverse Events and for laboratory assessments (v4.03) that include biochemistry, hematology, urinalysis; special safety assessments that include LVEF, Thyroid function Creatinine clearance and ECGs (electrocardiograms).

CONTACTS AND LOCATIONS:
Overall Officials: yue lu, MD., Principal Investigator — hematological oncology department
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No